CLINICAL TRIAL: NCT02034136
Title: Effects of Ginsenoside Supplementation on Insulin Resistance and Cardiometabolic Risk Factors in Men With Metabolic Syndrome: a Randomized Controlled Trial.
Brief Title: Ginsenoside Improve Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHA University (Other)
Collaborators: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Dong-Hyuk Jung, Assistant professor, Family medicine, CHA University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DH-13722; BD2013-104 (Other: Cha medical university IRB)
Record Dates: First submitted 2013-07-21; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Ginsenosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginsenoside (Experimental): Ginsenoside :
  Intervention : ginsenoside, 3 gram / day, for 28 days in intervention group
  Interventions: Dietary Supplement: Ginsenoside
- Dietary fiber fill (Placebo Comparator): Dietary fiber fill manufactured to mimic Ginsenoside tablet
  Interventions: Dietary Supplement: Dietary fiber fill

INTERVENTIONS:
Dietary Supplement: Ginsenoside — 3.0 g/ d for 28 days
  Other Names: Ginseng fill
  Arms: Ginsenoside
Dietary Supplement: Dietary fiber fill — 3g/day, 28days
  Arms: Dietary fiber fill

SUMMARY:
Aim : Investigated the effects of Korean red ginseng supplementation on metabolic parameters such as cholesterol, blood pressure and glucose.

Randomized Control Trial.

DETAILED DESCRIPTION:
Methods : A randomized, double-blind, placebo-controlled, single-center study in 60 subjects who are not taking drugs that could affect metabolic and vascular function. Subjects will be randomized into a Korean red ginseng (3.0g/d) group or placebo group for a 4-week study.

We will collect anthropometric measurements, blood for laboratory testing, inflammatory marker, hormones and mitochondrial DNA copy number.

Subject : Older than 40 years of age, presented with metabolic syndrome. Subjects were excluded if they were taking drugs that could affect metabolic and vascular function, including BP control drug, anti-diabetic drugs and lipid-lowering drugs.

Measurement : We will collect anthropometric measurements and blood for laboratory testing at the initial(week 0) and final (week 4)visits. Serum levels of blood glucose, insulin, total cholesterol, HDL-cholesterol,triglyceride, and DNA copy number of mitochondria.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome

Exclusion Criteria:

* Taking drug for lipid-lowering, BP control and anti-diabetic.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in metabolic syndrome profile at week 4 | Baseline and 4 weeks from intake of Ginsenoside
  Total cholesterol, HDL-Cholesterol, Glucose, Blood Pressure, Body weight

SECONDARY OUTCOMES:
Change from baseline in hormones at week 4. | Initial and 4 weeks later
  insulin ,cortisol, testosterone, somatomedin-c and DHEAS

OTHER OUTCOMES:
Mitochondria DNA copy number | initial and 4 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: DH Jung, MPH.M.D., Principal Investigator — Cha Medical University
Locations (1):
- Bundang CHA Hospital, Seoul, Kyeonggi-do, South Korea

REFERENCES:
- [Background] Park BJ, Lee YJ, Lee HR, Jung DH, Na HY, Kim HB, Shim JY. Effects of Korean Red Ginseng on Cardiovascular Risks in Subjects with Metabolic Syndrome: a Double-blind Randomized Controlled Study. Korean J Fam Med. 2012 Jul;33(4):190-6. doi: 10.4082/kjfm.2012.33.4.190. Epub 2012 Jul 25. PMID 22916320
- [Background] Rasheed N, Tyagi E, Ahmad A, Siripurapu KB, Lahiri S, Shukla R, Palit G. Involvement of monoamines and proinflammatory cytokines in mediating the anti-stress effects of Panax quinquefolium. J Ethnopharmacol. 2008 May 8;117(2):257-62. doi: 10.1016/j.jep.2008.01.035. Epub 2008 Feb 8. PMID 18339495
- [Background] Lamers F, Vogelzangs N, Merikangas KR, de Jonge P, Beekman AT, Penninx BW. Evidence for a differential role of HPA-axis function, inflammation and metabolic syndrome in melancholic versus atypical depression. Mol Psychiatry. 2013 Jun;18(6):692-9. doi: 10.1038/mp.2012.144. Epub 2012 Oct 23. PMID 23089630
- [Background] Yun SN, Ko SK, Lee KH, Chung SH. Vinegar-processed ginseng radix improves metabolic syndrome induced by a high fat diet in ICR mice. Arch Pharm Res. 2007 May;30(5):587-95. doi: 10.1007/BF02977653. PMID 17615678
- [Background] Kim JH, Lee DC. Mitochondrial DNA copy number in peripheral blood is associated with femoral neck bone mineral density in postmenopausal women. J Rheumatol. 2012 Jul;39(7):1465-72. doi: 10.3899/jrheum.111444. Epub 2012 May 15. PMID 22589267
- [Derived] Jung DH, Lee YJ, Kim CB, Kim JY, Shin SH, Park JK. Effects of ginseng on peripheral blood mitochondrial DNA copy number and hormones in men with metabolic syndrome: A randomized clinical and pilot study. Complement Ther Med. 2016 Feb;24:40-6. doi: 10.1016/j.ctim.2015.12.001. Epub 2015 Dec 4. PMID 26860800
- See also: The goal of Korean ginsengsociety is to help elevate the level of ginseng science in both theory and practice by providing technical information to the ginseng industry, providing ginseng-related education to the community. — http://www.ginsengsociety.org/